CLINICAL TRIAL: NCT05534997
Title: Effect of Intensive Combined Rehabilitation Therapy for Patients With Post COVID 19 Chronic Fatigue Syndrome
Brief Title: Rehabilitation Therapy for Post COVID 19 Chronic Fatigue Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Hosny, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chronic fatigue syndrome
Record Dates: First submitted 2022-08-26; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Post-COVID-19 Syndrome
Keywords: chronic fatigue; graded exercise; cognitive behavioral therapy
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: pre and post test parallel groups randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): will receive the post covid protocol conventional treatment in form of medication and 24 sessions of combined rehabilitation exercise program in the form of Graded exercise therapy (GET) and cognitive behavioral therapy (CBT). Patients will attend two sessions per week for 12 weeks. Sessions will be taken at Modern university for technology and information physical therapy rehabilitation center . A home exercise program will be prescribed on at least five days a week. Patients will be contacted by phone daily for the 12 weeks treatment sessions, for following up the home exercise program.
  Interventions: Other: intensive combined rehabilitation therapy
- Group B (No Intervention): will receive the post covid protocol conventional treatment in form of medication and specialist medical care provided by doctors with specialist experience in CFS. All patients will be given a leaflet explaining the illness and the nature of this treatment. Treatment will consist of an explanation of chronic fatigue syndrome, generic advice such as to avoid extremes of activity and rest, specific advice on self-help and symptomatic pharmacotherapy (especially for insomnia, pain and mood) .

INTERVENTIONS:
Other: intensive combined rehabilitation therapy — graded exercise therapy and cognitive behavioral therapy
  Arms: Group A

SUMMARY:
The aim of this study is to investigate the effect of intensive combined rehabilitation therapy in form of Graded Exercise Therapy (GET) , Cognitive Behavioral Therapy (CBT) to treat patients with post COVID19 chronic fatigue syndrome .

DETAILED DESCRIPTION:
A significant proportion of COVID-19 patients are suffering from prolonged Post-COVID-19 Fatigue Syndrome, with characteristics typically found in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). More recent studies of post-COVID-19 patients, over an extended period (6 months or more), have highlighted post-exertional malaise and relapses, both key characteristics of ME/CFS.

With over 147 million confirmed cases of COVID-19 worldwide currently and globally, the number of post-COVID-19 patients with chronic fatigue syndrome like symptoms is likely to be in the order of millions. This will present a worldwide, significant, ongoing health problem. With this impending flow of health crisis, it is hoped more intensive research into post covid chronic fatigue syndrome with a specific focus on study of these illnesses will likely bring significant advances.

Chronic fatigue syndrome is a disabling condition with a high impact on individuals and society, which causes a substantial economic burden. The persistent and debilitating nature of chronic fatigue syndrome often results in a reduction in work and family life activities, as well as an increase in health care costs. Because it becomes difficult for patients with chronic fatigue syndrome to continue employment at morbid levels, many have little choice but to leave their jobs.

Management of fatigue states requires multidisciplinary input and will not be appropriately addressed if follow-up is by treating medical physicians alone. A suite of interventions, including graded exercise and cognitive behavioral therapy, are needed to manage chronic fatigue syndrome and may be relevant to post infectious fatigue.

Research evaluating the efficacy of graded exercise therapy (GET) in alleviating the symptoms of chronic fatigue found that at the end of treatment, the exercise group rated themselves as significantly more improved and less fatigued than the control group. A decrease in symptom focusing rather than an increase in fitness mediated the treatment effect. Graded exercise appears to be an effective treatment for CFS, and it operates in part by reducing the degree to which patients focus on their symptoms.

Regarding several RCTs, a systematic review concluded that cognitive-behavioral therapy (CBT) interventions showed promising results, appearing to reduce fatigue and improve physical functioning. A Cochrane review on cognitive behavioral therapy in adults with chronic fatigue syndrome stated that cognitive-behavioral therapy (CBT) is effective in reducing the symptoms of fatigue at post treatment compared with usual care, and maybe more effective in reducing fatigue symptoms compared with other psychological therapies. Fifteen studies were included in the review. When comparing cognitive-behavioral therapy (CBT) with usual care, the difference in fatigue means scores at post treatment was highly significant in favor of that of cognitive-behavioral therapy (CBT) , with 40% of CBT showing clinical response in contrast with 26% in usual care.

A systematic review of randomized controlled trials of treatments for chronic fatigue syndrome found that graded exercise therapy (GET) and cognitive-behavioral therapy (CBT) are effective for patients with chronic fatigue syndrome, the overall results of studies suggested a significant positive effect on fatigue, symptoms and improvements in measures of physical function. Graded exercise works best for chronic fatigue syndrome (CFS) when combined with cognitive-behavioral therapy (CBT).

Training studies of High-intensity interval training (HIIT) have revealed more favorable results in a variety of physiological outcomes when compared with traditional continuous training . High-intensity interval training (HIIT) has been shown to be safe and to produce improvements in quality of life . Participants have also reported HIIT to be more enjoyable than moderate-intensity continuous training .

Previous studies have indicated that high-intensity interval training (HIIT) was an effective exercise for the enhancement of aerobic and anaerobic capacity . This phenomenon is attributed to increases in the heart's pumping capacity and the mitochondrial activity . Increased aerobic capacity is related to health benefits such as longer lifespan, functional independence, psychological well-being, and quality of life .

High-intensity interval training ( HIIT) appears to be a safe and well-tolerated supplement to proven fall prevention programs, due to its effects on lower limb strength reflected in functional performance tests, and on dynamic balance and subjective balance perception . So high-intensity interval training ( HIIT) will be included, as part of Graded exercise therapy GET in our study. No available research work investigates the effect of Cognitive Behavioral Therapy (CBT) and graded exercise therapy (GET) on post COVID-19 chronic fatigue syndrome.

So the aim of this study is to investigate the effect of intensive combined rehabilitation therapy in form of Graded Exercise Therapy (GET) , Cognitive Behavioral Therapy (CBT) to treat patients with post COVID-19 chronic fatigue syndrome .

ELIGIBILITY:
Inclusion Criteria:

* 60 post covid patients (6 months recovery after last negative PCR diagnosis)
* Patients will be selected using the Oxford diagnostic criteria for CFS which required disabling fatigue to be the primary problem, in the absence of an exclusionary medical or psychiatric diagnosis. Patients will fulfil the following criteria for CFS :

  * fatigue as a principal symptom.
  * fatigue definite onset that is not life long.
  * fatigue should have been present for a minimum of 6 months during which it was present for more than 50% of the time.
  * Other symptoms may be present, particularly myalgia, mood and sleep disturbance.
* Both sexs will be included
* Body mass index range from (18.5 to 24.9 kg/m2)
* Patients' age range will be 18 to 34 years old .
* Presence of significant fatigue since COVID-19.
* Able to understand and willing to sign a written informed consent document.
* Willing and able to complete study procedures.

Exclusion Criteria:

* On medications that would influence exercise performance such as beta blockers or antiretroviral therapy
* Enrolled in another interventional clinical research trial
* Pregnancy
* Significant hepatic or renal dysfunction
* History or cardiac condition as determined by National Institutes of Health (NIH) cardiology to be unsafe for exercise participation (e.g. ischemic heart disease, right- or left-sided heart failure, cor pulmonale or pulmonary hypertension, dilated or hypertrophic cardiomyopathy or non-idiopathic cardiomyopathy)
* Patients with a current diagnosis of schizophrenia, manic depressive illness, substance abuse, eating disorder or proven organic brain disease.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The fatigue severity level | 12 weeks
  The fatigue severity level will be measured via the Arabic version of the Fatigue Severity Scale (FSS)
aerobic capacity and endurance | 12 weeks
  Aerobic capacity and endurance will be measured via The 6 Minute Walk Test. The test will be performed at Modern University for the technology and information rehabilitation center corridor.
Maximal hand grip strength and fatigue resistance | 12 weeks
  Maximal hand grip strength and fatigue resistance will be measured using the Handgrip dynamometer
the Fall risk | 12 weeks
  Fall risk will measure via the Biodex Balance System (BBS) (Biodex Medical Systems Inc, Shirley, NY).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenhalgh T, Knight M, A'Court C, Buxton M, Husain L. Management of post-acute covid-19 in primary care. BMJ. 2020 Aug 11;370:m3026. doi: 10.1136/bmj.m3026. No abstract available. PMID 32784198
- [Background] Elboim-Gabyzon M, Buxbaum R, Klein R. The Effects of High-Intensity Interval Training (HIIT) on Fall Risk Factors in Healthy Older Adults: A Systematic Review. Int J Environ Res Public Health. 2021 Nov 11;18(22):11809. doi: 10.3390/ijerph182211809. PMID 34831565
- [Background] Dennis A, Wamil M, Alberts J, Oben J, Cuthbertson DJ, Wootton D, Crooks M, Gabbay M, Brady M, Hishmeh L, Attree E, Heightman M, Banerjee R, Banerjee A; COVERSCAN study investigators. Multiorgan impairment in low-risk individuals with post-COVID-19 syndrome: a prospective, community-based study. BMJ Open. 2021 Mar 30;11(3):e048391. doi: 10.1136/bmjopen-2020-048391. PMID 33785495
- [Background] Deale A, Chalder T, Marks I, Wessely S. Cognitive behavior therapy for chronic fatigue syndrome: a randomized controlled trial. Am J Psychiatry. 1997 Mar;154(3):408-14. doi: 10.1176/ajp.154.3.408. PMID 9054791